CLINICAL TRIAL: NCT06972654
Title: Efficacy of Combined Nalbuphine-bupivacaine Versus Dexamethasone-bupivacaine in Pericapsular Nerve Group Block (PENG) for Postoperative Analgesia in Hip Surgeries: A Randomized Clinical Study
Brief Title: Analgesic Effects of Combined Nalbuphine-bupivacaine Versus Dexamethasone-bupivacaine in Pericapsular Nerve Group Block (PENG) After Hip Surgeries: A Randomized Clinical Study
Acronym: PENG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Abdelhameed Elsadek Salem, PRINCIPLE INVESTIGATOR, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1112
Record Dates: First submitted 2025-03-25; First posted 2025-05-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-03

CONDITIONS: Analgesia, Postoperative
Keywords: nalbuphine-bupivacaine; ultrasound guided pericapsular nerve group (PENG); dexamethasone-bupivacaine
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Evaluate the efficacy of nalbuphine-bupivacaine vs dexamethasone-bupivacaine in ultrasound guided pericapsular nerve group (PENG) block for improving pain management, reducing opioid consumption, and enhancing the overall analgesic effect in patients undergoing hip surgeries
Who Masked: Participant, Outcomes Assessor
Masking Description: Anesthetist not sharing in the study will assess patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Bupivacaine + nalbuphine (N) (Active Comparator): Patients in this group will receive a unilateral ultrasound-guided pericapsular nerve group (PENG) block with a combination of 20 mL of bupivacaine 0.25%- and 2 ml nalbuphine (20 mg), with total volume 22ml
  Interventions: Procedure: Group Nalupnine
- Group Bupivacaine + dexamethasone (D) (Active Comparator): Patients in this group will receive a unilateral ultrasound-guided PENG block with a combination of 20 mL of bupivacaine 0.25%- , 1 ml dexamethasone (4 mg) and 1 ml saline, with total volume 22ml
  Interventions: Procedure: Group Dexamethasone

INTERVENTIONS:
Procedure: Group Nalupnine — Patients will receive a unilateral ultrasound-guided pericapsular nerve group (PENG) block with a combination of 20 mL of bupivacaine 0.25%- and 2 ml nalbuphine (20 mg), with total volume 22ml.
  Arms: Group Bupivacaine + nalbuphine (N)
Procedure: Group Dexamethasone — Patients will receive a unilateral ultrasound-guided PENG block with a combination of 20 mL of bupivacaine 0.25%- 1 ml dexamethasone (4 mg) and 1 ml saline, with total volume 22ml
  Arms: Group Bupivacaine + dexamethasone (D)

SUMMARY:
The aim of the study to Evaluate the efficacy of nalbuphine-bupivacaine vs dexamethasone-bupivacaine in ultrasound guided pericapsular nerve group (PENG) block for improving pain management, reducing opioid consumption, and enhancing the overall analgesic effect in patients undergoing hip surgeries.

DETAILED DESCRIPTION:
1. To measure the time of first request of rescue analgesia , the total amount of rescue analgesic consumption (pethidine) in the first 24 hours post-operatively in each group and number of patients received one or two doses rescue analgesia.
2. To assess pain score by using numerical rate scale (NRS) at rest (static) and during passive flexion or extension of hip (dynamic).
3. To assess the incidence of drug-related side effects (such as nausea, vomiting, bradycardia, hypotension, sedation and hyperglycemia) or block -related side effects (hematoma, infection or LA toxicity) in patients receiving either nalbuphine or dexamethasone as adjuvant to bupivacaine in the PENG block.
4. To assess Ease of Spinal Positioning (EOSP).
5. To assess patient satisfaction.

ELIGIBILITY:
Inclusion criteria:

* Patients acceptance.
* Age: Adults aged 21-75 years old.
* BMI: 25-30 kg/m2
* Sex: both sexes (males or females).
* Patients undergoing unilateral hip surgery under spinal anesthesia.
* ASA (American Society of Anesthesiologists) physical status classification I, II and Ⅲ..

  *Exclusion criteria:
* Patients with contraindications to regional anesthesia (e.g. local or systemic infections, or severe neurological or muscular disorders or patient on anticoagulant).
* Allergy to study drugs: bupivacaine or nalbuphine or dexamethasone
* Patients with severe cardiovascular, respiratory, renal, or hepatic conditions, uncontrolled diabetes diseases, or those undergoing chronic opioid therapy.
* Psychiatric disorders that hinder informed consent or study participation.
* history of neurological diseases or conditions that would affect the efficacy of nerve blocks (e.g., neuropathy, spinal cord injury, or history of severe muscle weakness).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
The time to first request of rescue analgesia | 24 hours postoperative
  (time from end of local anesthetics injection in PENG block till time of NRS >3) will be recorded.

SECONDARY OUTCOMES:
postoperative pain by Numerical Rating Scale | Basal (before giving the block), 15 minutes after giving the block and before spinal anesthesia, PACU ( after arrival to PACU 0 minute), 2 hours (hrs), 4 hrs, 8 hrs, 12 hrs and 24 hrs.
  To assess pain score by using numerical rate scale (NRS) at rest (static) and during passive flexion or extension of hip (dynamic) at different time points
To assess the total amount of rescue analgesic consumption | 24 hours postoperative
  To assess the total amount of rescue analgesic consumption in the first 24 hours post-operatively in each group
To assess the incidence of drug-related side effects or block -related side effects | 24 hours postoperative
  To assess the incidence of drug-related side effects (such as nausea, vomiting, respiratory depression and hyperglycemia) or block -related side effects (hematoma, infection or LA toxicity) in patients receiving either nalbuphine or dexamethasone as adjuvant to bupivacaine in the PENG block.
Ease of Spinal Positioning (EOSP) | up to 15 minutes after giving the block
  evaluated on a scale from zero to three (zero = unable to be positioned; one = abnormal posture of the patient due to pain requiring support for positioning; two = mild discomfort but no need for assisted positioning; three = optimal condition where the patient could sit without feeling pain)
patient's satisfaction | 24 hours postoperative
  overall degree of satisfaction of the analgesia by using a 5-points Likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia)
Number of patients received one or two doses rescue analgesia | 24 hours
  Number of patients received one or two doses rescue analgesia (pethidine) postoperative
Length of hospital stay | up to 5 days
  number of hospital stay days starting from PACU discharge till home discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Faculity of medicine, Zagazig university, Zagazig, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No